CLINICAL TRIAL: NCT05618067
Title: The Impact of Improved Vagal Function on Periaqueductal Gray Connectivity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20025315
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental)
  Interventions: Behavioral: breathing exercise training

INTERVENTIONS:
Behavioral: breathing exercise training — Participants will engage in weekly breathing exercises. They will be trained once a week for 4 weeks, and will use an app called Inner Balance and an device called Firstbeat Bodyguard 3 to track data about their hearts while practicing the exercises at home for 10 minutes a day, twice a day, once before bedtime.

SUMMARY:
This study is being to see if participating in breathing exercise training and practicing this training will help with Postural tachycardia syndrome (POTS). The information may help doctors to learn more about how the different parts of people's brains communicate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Diagnosis of POTS, orthostatic intolerance (with or without syncope), syncope, or near-syncope
* Can speak and read in English
* Upcoming new patient VCU Comprehensive Autonomics Center clinic visit scheduled at least 1 week in the future

Exclusion Criteria:

* Inflammatory arthritis, connective tissue or auto-immune disorder
* Any chronic neurological disorder besides POTS, orthostatic intolerance (with or without syncope), syncope, or near-syncope
* Patients who have already had a new patient clinic visit where they were exposed to breathing exercise education
* Evidence of unstable medical disorder, such as kidney (rising creatinine, or end-stage renal failure) or liver impairment (rising AST or ALT, or end-stage with coagulopathy), poorly controlled significant cardiovascular (CHF), respiratory, endocrine (diabetes - A1c > 9 - or untreated thyroid dysfunction) or uncontrolled psychiatric illness (such as untreated depression, psychosis, etc.)
* Neuropathy, central nervous system disorder (e.g., Cerebral palsy, developmental delay, seizure disorder, MS, stroke, etc.)
* Treatment with a drug or medical device within the previous 30 days that has not received regulatory approval
* Use of hormones (except insulin, thyroid replacement or oral contraceptives, which will be carefully documented)
* Current substance or alcohol abuse
* Any major surgical intervention with general anesthesia in the last 60 days and minor procedure, such as tooth extraction, endoscopy, etc., with local or conscious sedation within 7 days
* Any on-going or pending medical, health or disability related litigation, or current pursuit of disability
* Any condition that in the judgment of the investigator would interfere with the patient's ability to provide informed consent, comply with study instructions, place the patient at increased risk, or which would clearly confound the interpretation of the study results (specific reason will be documented)
* Chronic use of narcotics for pain
* Claustrophobia or any metal hardware that may interfere with MRI
* Investigators and study staff

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in periaqueductal gray region (PAG) activation - looming task | 90 minutes
  Functional magnetic resonance imaging (fMRI) will be performed to measure activation of the PAG region during the looming task
Change in PAG activation - resting | 90 minutes
  Functional magnetic resonance imaging (fMRI) will be performed to measure activation of the PAG region while at rest
Change in Heart Rate Variability (HRV) | Assessed for 2 days each week for the duration of the study (6 weeks).
  HRV will be measured using an ear clip and/or wristband and results will be recorded automatically in the app

SECONDARY OUTCOMES:
Change in Fatigue Severity Scale (FSS) score from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue by asking participants to answer 9 statements that rate the severity of their fatigue symptoms in the past week by selecting their answer on a 1-7 point Likert scale. Sum scores range from 9-36. A low value (e.g., 1) indicates strong disagreement with the statement (lower symptom severity), whereas a high value (e.g., 7) indicates strong agreement (higher symptom severity).
Change in Generalized Anxiety Disorder Scale (GAD-2) score from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The Generalized Anxiety Disorder Scale (GAD-2) is a method of evaluating anxiety symptoms by asking participants to answer 2 statements that rate the severity of their anxiety symptoms in the past 2 weeks by selecting their answer a 0-3 point Likert scale (0- not at all, 1- several days, 2 - more than half the days, 3 - nearly every day). Sum scores range from 0-6. A low value (e.g., 0) indicates no or less severe anxiety symptoms, whereas a high value (e.g. 3), indicates more severe anxiety symptoms.
Differences in Adverse Childhood Experiences (ACE) scores between participants | Assessed at baseline.
  The Adverse Childhood Experiences (ACE) questionnaire is a method of evaluating childhood adversities such as emotional, physical, and sexual abuse/neglect by asking participants to answer 10 statements that describe events that happened during the first 18 years of their life. Participants indicate if this event occurred by selecting a Yes or No answer. Sum scores range from 0-10. Less "Yes" responses indicate less ACE occurrences, and more "Yes" responses indicate more ACE occurrences.
Change in Pain Catastrophizing Scale (PCS) score from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The Pain Catastrophizing Scale (PCS) is a method of evaluating pain catastrophizing, measuring pain-related cognitions and the dimensions of helplessness, rumination and magnification by asking participants to answer 13 items that describe different thoughts and feelings that may be associated with their pain. Participants rate how strong their feelings are about pain on a 5 point scale (0- Not at all, 1- To a slight degree, 2- To a moderate degree, 3- To a great degree, 4- All the time). Sum scores range from 0-52. Higher scores indicate higher levels of pain catastrophizing. A total PCS score of 30 represents a clinically relevant level of catastrophizing.
Change in Patient Health Questionnaire (PHQ-9) score from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The Patient Health Questionnaire (PHQ-9) objectifies and assesses degree of depression severity via questionnaire by asking participants to answer 9 items that rate the severity of depression symptoms over the past 2 weeks on a 0-3 point Likert scale (0- not at all, 1- several days, 2 - more than half the days, 3 - nearly every day). Sum scores range from 0-36. A low value (e.g., 0) indicates no or less severe depression symptoms, whereas a high value (e.g. 3), indicates more severe depression symptoms.
Change in Pittsburgh Sleep Quality Index (PSQI) from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The Pittsburgh Sleep Quality Index (PSQI) measures quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the past month. Participants are asked to answer 19 items. 5 items are free response and ask questions about sleep duration. The remaining 14 items are answered on a 0-3 point Likert scale (0 - not during the past month, 1- less than once a week, 2- once or twice a week, 3- three or more times a week) that describe the frequency of the listed events. A global score is calculated from the sum of 7 component scores and ranges from 0-21, with lower scores indicating lower sleep dysfunction and higher scores indicating higher sleep dysfunction.
Change in PROMIS Physical Function (PROMIS 8b) from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The PROMIS Physical Function (PROMIS 8b) instrument measures self-reported capability of physical activities by asking participants to respond to 8 items on a 5-point Likert scale. The scale for the first 4 items is as follows: 5- Without any difficulty, 4- With a little difficulty, 3- With some difficulty, 2- With much difficulty, 1- Unable to do. The scale for the last 4 items is as follows: 5- Not at all, 4- Very little, 3- Somewhat, 2- Quite a lot, 1- Cannot do. Raw sum scores range from 8-40 and are converted into a T-score ranging from 20.3 to 60.1, with higher scores indicating better physical function and lower scores indicating poorer physical function.
Change in the Perceived Stress Scale (PSS) from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The Perceived Stress Scale (PSS) measures how different situations affect feelings and perceived stress. Participants are asked to answer 10 items that describe the frequency of their feelings and thoughts described in each item during the last month on a 0-4 point Likert scale (0 - never, 1- almost never, 2- sometimes, 3- fairly often, 4- very often). Sum scores range from 0-40, with lower scores indicating less perceived stress levels and higher scores indicating higher perceived stress levels.
Change in the PTSD Checklist (PCL-5) from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The PCL-5 assesses the 20 DSM-5 symptoms of PTSD. Participants are asked to answer 5 free response questions about the worst & more stressful event to which they were exposed, then 20 items about the event on a 0-4 point Likert scale (0- not at all, 1- a little bit, 2- moderately, 3- quite a bit, 4- extremely). Sum scores of the 20 Likert-format items range from 0-80, with lower scores indicating less severe PTSD symptoms and higher scores indicating more severe PTSD symptoms.
Change in the Pain, Enjoyment of Life, and General Activity (PEG-3) from baseline | Assessed at baseline, week 3, and week 6 (final visit).
  The Pain, Enjoyment of Life, and General Activity (PEG-3) scale assesses pain levels and interference with enjoyment of life and activity. Participants are asked to answer 3 items on a 0-10 point Likert scale. For item 1, the scale is as follows: 0- no pain, 10- pain as bad as you can imagine. For items 2-3, the scale is as follows: 0- does not interfere, 10- completely interferes. Sum scores range from 0-30, with lower scores indicating less pain and/or interference and higher scores indicating more pain and/or interference.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chelimsky, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virnigia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No